CLINICAL TRIAL: NCT03044028
Title: Prospective Evaluation of Neuromuscular Electrical Stimulation (NMES) for Improving Outcomes Following Total Knee Arthroplasty (TKA)
Brief Title: Neuromuscular Electrical Stimulation (NMES) for Improving Outcomes Following Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Carlos Higuera-Rueda, Staff Surgeon, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #16-1293
Record Dates: First submitted 2016-12-20; First posted 2017-02-06 (Estimated); Results first posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Arthropathy of Knee Joint

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NMES preoperative and postoperative (Experimental): Subject will be given NMES CyMedica Orthopedics QB1 e-vive™ system device to use preoperative and will continue to use postoperatively until end of study
  Interventions: Device: CyMedica Orthopedics QB1 e-vive™ system
- NMES postoperative only (Experimental): Subject will be given NMES CyMedica Orthopedics QB1 e-vive™ system device to use postoperatively and will continue to use until end of study
  Interventions: Device: CyMedica Orthopedics QB1 e-vive™ system
- No intervention (No Intervention): Subject will not be given device and will undergo the standard rehab protocol alone

INTERVENTIONS:
Device: CyMedica Orthopedics QB1 e-vive™ system — a multifunctional electrotherapy device providing neuromuscular electrical stimulation (NMES), for improving quadriceps strength and improving functional outcomes accelerating functional recovery in patients managed with total knee arthroplasty (TKA).
  Other Names: NMES Neuromuscular electrical stimulation
  Arms: NMES postoperative only; NMES preoperative and postoperative

SUMMARY:
The current standard for rehabilitation after TKA consists of guided exercise therapy for up to 12 weeks after surgery. This includes inpatient, home, and outpatient therapy. The surgery and rehabilitation are highly successful at reducing or eliminating pain experienced preoperatively. However, quadriceps femoris muscle (QFM) strength, overall function, and knee range of motion are often worse than preoperative levels for as long as 6 months after surgery and in some cases may persist for many years after that. Such quadriceps strength impairments after TKA have been largely attributed to voluntary activation deficits and can lead to a decrease in functional performance such as decreased gait speed, decreased balance which can lead to falls, and decreased stair climbing & chair rise abilities.

Since therapy alone does not adequately restore or improve upon the preoperative functional capabilities in a consistent and timely manner, it has been suggested that NMES used adjunctively with postoperative rehabilitation will alleviate the quadriceps muscle activation deficits. Early NMES use after TKA has been shown to: reduce knee extensor lag, increase walking speed, and improve QFM strength, knee range of motion, and function. However, NMES initiated one month after TKA did not lead to improved QFM strength or function beyond the standard benefits gained from exercise alone, thus suggesting that the timing of NMES application after TKA is important.

It has previously been shown that preoperative QFM strength is predictive of postoperative function [6] but the benefit of prehabilitation remains in question. To date, there has only been one pilot study assessing the benefits of NMES when initiated preoperatively. This study only included 14 patients (9 NMES, 5 control) but was able to show that preoperative NMES usage may lead to greater QFM strength gains after TKA. Therefore, it will be important to assess the benefits of NMES both preoperatively and postoperatively in order to determine how it will be most beneficial to TKA patients.

DETAILED DESCRIPTION:
The study duration will be until 12 weeks ± 1 week postoperatively. Data will be collected (1) 4 weeks preoperatively, (2) prior to hospital admission for TKA, and (3) at 3, 6, and 12 weeks postoperatively. The research coordinator at the site will identify, recruit, and prospectively follow the 66 patients at his/her site.

All data will be entered and maintained in REDCap, an electronic data capture tools hosted at Cleveland Clinic. REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies, providing 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources. Only members of the study team (i.e. the personnel listed on the institutional review board (IRB) application) will have access to protected health information of patients included in this study.

Pretreatment Assessments

Before treatment, the following assessments/tests will be performed and the results will be recorded on the appropriate pages of the (case report form) CRF, and or Microsoft excel, Microsoft Word, and REDCap:

* Informed consent
* Age, gender, height/weight/(body mass index) BMI
* Concomitant diseases
* Physical examination
* Baseline range of motion of affected knee
* Baseline timed up and go test (TUG test, detailed in Appendix A and as described by Podsiadlo et al.)
* Baseline Stair Climb test
* Baseline QFM strength
* Baseline Modified Knee Injury and Osteoarthritis Outcome Score (KOOS) and Veterans Rand 12(VR-12) assessments
* Baseline VAS (visual analog scale)pain score
* Current medications
* Any use of ambulation assist device

Presurgery Assessments

Before surgery, the following assessments/tests will be performed and the results will be recorded on the appropriate pages of the CRF, and or Microsoft excel, Microsoft Word, and REDCap:

* Device usage patterns (thru app for preop NMES group)
* Range of motion of affected knee
* TUG test
* Stair Climb test
* QFM strength
* Modified KOOS and VR-12 assessments
* VAS pain score
* Current medications
* Activity levels using Misfit Wearables® fitness monitor will be uploaded and incorporated into online app

Operative Assessments

The following will be collected from the Operative and Anesthesia Records and recorded on the appropriate pages of the CRF, and or Microsoft excel, Microsoft Word, and REDCap:

* Surgeon name
* Approach used
* Randomization assignment
* Diagnosis
* Length of surgery
* Estimated blood loss
* Type of anesthesia
* Implant type

Postoperative Assessments After surgery, one or more of the following will be collected through the online app and at follow-up visits.

* Device usage patterns (thru app)
* Range of motion of affected knee (thru app and at follow-up)
* TUG test
* Stair Climb test
* QFM strength
* Modified KOOS and VR-12 assessments
* VAS pain score
* Length of stay (hospital, extended care facility)
* 90 day readmission rate
* Discharge Disposition (home vs skilled nursing facility vs inpatient rehabilitation)
* Patient Satisfaction measures
* Any use of an ambulation assist aid
* Activity levels using Misfit Wearables® fitness monitor will be uploaded and incorporated into online app

As a last resort, if a patient is unable to keep one of these appointments, he/she will be either be mailed or emailed the patient reported outcome forms so the patient can fill them out. The patient will date and time the forms. Participants will then send the form back in a pre-addressed envelope. The patients email will be verified by the patient during a clinical visit to ensure accuracy of the correct recipient. Patients not responding to the initial mailer will be contacted by phone and forms may be administered over the phone. The mailers and/or phone calls will allow us to collect all data except the physical function measures.

All data will be entered and maintained in Redcap

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing unilateral primary total knee arthroplasty
2. Patients who are between the ages of 18 - 85 years
3. Patient has signed informed consent
4. Patient has access to a smartphone or tablet (Android or iOS)

Exclusion Criteria:

1. BMI ≥ 40
2. Inflammatory arthritis
3. Patients who are expected to be in extended care facilities after surgery
4. Patients who have used an at-home NMES device in the past
5. Preoperative daily use of narcotics (i.e., high tolerance)
6. Already enrolled in another research study, including the present study for contralateral knee
7. Other lower-extremity orthopaedic conditions which could interfere with limb function, especially those with significant pain requiring daily analgesic intake
8. Patients with concurrent abdominal, inguinal or femoral hernias
9. Cutaneous lesions in areas of electrode pad placement
10. Patients with a history of epilepsy
11. Patients with a cardiac pacemaker/defibrillator
12. Allergy to adhesives
13. Inability to meet follow-up visits required for the study
14. Patients who are a risk for poor compliance or have a poor understanding of the use of the NMES device
15. Condition deemed by physician or medical staff to be non-conducive to patient's ability to complete the study, or a potential risk to the patient's health and well-being

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01; Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mont, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stevens-Lapsley JE, Balter JE, Wolfe P, Eckhoff DG, Kohrt WM. Early neuromuscular electrical stimulation to improve quadriceps muscle strength after total knee arthroplasty: a randomized controlled trial. Phys Ther. 2012 Feb;92(2):210-26. doi: 10.2522/ptj.20110124. Epub 2011 Nov 17. PMID 22095207
- [Background] Levine M, McElroy K, Stakich V, Cicco J. Comparing conventional physical therapy rehabilitation with neuromuscular electrical stimulation after TKA. Orthopedics. 2013 Mar;36(3):e319-24. doi: 10.3928/01477447-20130222-20. PMID 23464951
- [Background] Gotlin RS, Hershkowitz S, Juris PM, Gonzalez EG, Scott WN, Insall JN. Electrical stimulation effect on extensor lag and length of hospital stay after total knee arthroplasty. Arch Phys Med Rehabil. 1994 Sep;75(9):957-9. PMID 8085929
- [Background] Avramidis K, Karachalios T, Popotonasios K, Sacorafas D, Papathanasiades AA, Malizos KN. Does electric stimulation of the vastus medialis muscle influence rehabilitation after total knee replacement? Orthopedics. 2011 Mar 11;34(3):175. doi: 10.3928/01477447-20110124-06. PMID 21410130
- [Background] Petterson SC, Mizner RL, Stevens JE, Raisis L, Bodenstab A, Newcomb W, Snyder-Mackler L. Improved function from progressive strengthening interventions after total knee arthroplasty: a randomized clinical trial with an imbedded prospective cohort. Arthritis Rheum. 2009 Feb 15;61(2):174-83. doi: 10.1002/art.24167. PMID 19177542
- [Background] Mizner RL, Petterson SC, Stevens JE, Axe MJ, Snyder-Mackler L. Preoperative quadriceps strength predicts functional ability one year after total knee arthroplasty. J Rheumatol. 2005 Aug;32(8):1533-9. PMID 16078331
- [Background] D'Lima DD, Colwell CW Jr, Morris BA, Hardwick ME, Kozin F. The effect of preoperative exercise on total knee replacement outcomes. Clin Orthop Relat Res. 1996 May;(326):174-82. doi: 10.1097/00003086-199605000-00020. PMID 8620638
- [Background] Villadsen A. Neuromuscular exercise prior to joint arthroplasty in patients with osteoarthritis of the hip or knee. Dan Med J. 2016 Apr;63(4):B5235. No abstract available. PMID 27034190
- [Background] Rodgers JA, Garvin KL, Walker CW, Morford D, Urban J, Bedard J. Preoperative physical therapy in primary total knee arthroplasty. J Arthroplasty. 1998 Jun;13(4):414-21. doi: 10.1016/s0883-5403(98)90007-9. PMID 9645522
- [Background] Walls RJ, McHugh G, O'Gorman DJ, Moyna NM, O'Byrne JM. Effects of preoperative neuromuscular electrical stimulation on quadriceps strength and functional recovery in total knee arthroplasty. A pilot study. BMC Musculoskelet Disord. 2010 Jun 14;11:119. doi: 10.1186/1471-2474-11-119. PMID 20540807
- [Background] Klika AK, Gehrig M, Boukis L, Milidonis MK, Smith DA, Murray TG, Barsoum WK. A Rapid Recovery Program After Total Knee Arthroplasty. Semin Arthro. 2009; 20:40-44.
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Brazier JE, Roberts J. The estimation of a preference-based measure of health from the SF-12. Med Care. 2004 Sep;42(9):851-9. doi: 10.1097/01.mlr.0000135827.18610.0d. PMID 15319610
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | No Intervention
Started | 22 | 22 | 22
Completed | 12 | 12 | 22
Not Completed | 10 | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | No Intervention | Total
Number analyzed (Participants) | 12 | 12 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (5.2) | 66.6 (6.3) | 64.5 (7.6) | 64.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 17 | 35
  Male | 3 | 3 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race not collected
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Femoris Muscle (QFM) Strength (Dynamometer Quad Strength Lbs)
Description: measure change in muscle strength (QFM) - difference from baseline measure to 6 weeks postoperative
Time Frame: 6 weeks
Population: Numbers do not match Participant Flow because data were missing.
Measure: Mean (Standard Deviation); unit: lbs
Groups:
- NMES Preoperative and Postoperative: NMES Preoperative and Postoperative, patients used the device a minimum of 900 minutes total preoperatively, and 200 min/wk postoperatively
- NMES Postoperative Only: NMES Postoperative only, patients used the device a minimum of 200 min/wk postoperatively
- Control - no NMES: Control - no NMES, patients did not use the device
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | Control - no NMES
Number analyzed (Participants) | 11 | 10 | 16
lbs | 3.35 (20.70) | 15.95 (14.61) | -5.48 (16.53)

2. Secondary Outcome: Knee Active Range of Motion (Extension, Flexion) in Degrees
Description: Measure rage of motion differences between the treatment groups
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | Control - no NMES
Number analyzed (Participants) | 12 | 12 | 22
degrees | 0.50 (13.22) | 6.67 (15.40) | -1.50 (12.93)

3. Secondary Outcome: Visual Analogue Scale (VAS) Pain Level (0-10 Scale)
Description: Differences in VAS scores between the treatment groups from baseline to 12 weeks postop. Higher score represents worse pain.
Time Frame: 12 weeks
Population: Numbers do not match Participant Flow because data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | Control - no NMES
Number analyzed (Participants) | 12 | 10 | 22
units on a scale | 2.00 (2.92) | 1.80 (2.04) | 1.18 (2.36)

4. Secondary Outcome: Hospital Length of Stay (Days)
Description: differences in length of stay between the treatment groups
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | Control - no NMES
Number analyzed (Participants) | 12 | 12 | 22
days | 1.83 (0.72) | 1.75 (0.45) | 1.68 (0.78)

5. Secondary Outcome: Number of Patients Discharged to Extended Care Facility
Description: Patent discharge other than "home" to extended care facility
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- NMES Postoperative Only: NMES Postoperative only, patients used the device a minimum 200 min/wk postoperatively
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | Control - no NMES
Number analyzed (Participants) | 12 | 12 | 22
Participants | 0 | 0 | 1

6. Secondary Outcome: Number of Patients Readmitted to Hospital
Description: Number of all-cause readmissions to the hospital
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | Control - no NMES
Number analyzed (Participants) | 12 | 12 | 22
Participants | 0 | 0 | 1

7. Secondary Outcome: Number of Outpatient Therapy Visits (Patient Questionnaire)
Description: Difference in number of outpatient therapy visits among the treatment groups
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | Control - no NMES
Number analyzed (Participants) | 7 | 8 | 21
visits | 12.86 (4.95) | 16.25 (7.29) | 11.67 (5.06)

8. Secondary Outcome: KOOS - PS
Description: Functional outcomes using the Knee Injury and Osteoarthritis Outcome Score (KOOS) Physical Function Shortform (PS) questionnaire. Change in total score from baseline to 12 weeks postoperative score. Minimum value is 0, maximum value is 100, and higher values mean greater improvement over baseline total score.
Time Frame: 12 weeks
Population: Numbers do not match Participant Flow because data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | Control - no NMES
Number analyzed (Participants) | 9 | 10 | 16
units on a scale | 33.43 (14.76) | 20.39 (12.70) | 26.62 (9.81)

9. Secondary Outcome: KOOS Pain
Description: Measure pain at 12 weeks postoperative using Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain subscore. Change in total score from baseline to 12 weeks postoperative score. Minimum value is 0, maximum value is 100, and higher values mean greater improvement over baseline total score.
Time Frame: 12 weeks
Population: Numbers do not match Participant Flow because data were missing.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | Control - no NMES
Number analyzed (Participants) | 9 | 10 | 16
z-score | 72.22 (19.64) | 78.89 (16.57) | 80.38 (15.43)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through 12 weeks postoperative.
Arm/Group | NMES Preoperative and Postoperative | NMES Postoperative Only | Control - no NMES
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NMES Preoperative and Postoperative (N=22) | NMES Postoperative Only (N=22) | Control - no NMES (N=22)
Readmission (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Patient was having abdominal pain and was admitted to hospital. Problem unrelated to study and resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT03044028/Prot_SAP_000.pdf